CLINICAL TRIAL: NCT02935855
Title: Efficacy and Safety of Non-vitamin K Oral Anticoagulants and Vitamin K Oral Anticoagulants on Some Metabolic and Coagulation Parameters in Diabetic and Nondiabetic Patients With First Diagnosis of Non-valvular Atrial Fibrillation
Brief Title: ORal anticoaGulants in diAbetic and Nondiabetic Patients With nOn-valvular Atrial fibrillatioN (ORGANON)
Acronym: ORGANON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20150003862
Record Dates: First submitted 2016-10-01; First posted 2016-10-18 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Diabetes
Keywords: Diabetic patients; nondiabetic patients
MeSH Terms: conditions — Diabetes Mellitus | interventions — Dabigatran; apixaban; Rivaroxaban; edoxaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nondiabetics (group 1) (Active Comparator): Nondiabetic patients with first diagnosis of non-valvular atrial fibrillation; they will be treated with dabigatran or apixaban or rivaroxaban or edoxaban in randomized way
  Interventions: Drug: Dabigatran; Drug: Apixaban; Drug: Rivaroxaban; Drug: Edoxaban
- Diabetics (group 1) (Active Comparator): Diabetic patients with first diagnosis of non-valvular atrial fibrillation; they will be treated with dabigatran or apixaban or rivaroxaban or edoxaban in randomized way
  Interventions: Drug: Dabigatran; Drug: Apixaban; Drug: Rivaroxaban; Drug: Edoxaban
- Nondiabetics (group 2) (Active Comparator): Nondiabetic patients with first diagnosis of non-valvular atrial fibrillation; they will be treated with warfarin or acenocumarole as guidelines suggest
  Interventions: Drug: Warfarin; Drug: Acenocumarole
- Diabetics (group 2) (Active Comparator): Diabetic patients with first diagnosis of non-valvular atrial fibrillation; they will be treated with warfarin or acenocumarole as guidelines suggest
  Interventions: Drug: Warfarin; Drug: Acenocumarole

INTERVENTIONS:
Drug: Dabigatran
  Arms: Diabetics (group 1); Nondiabetics (group 1)
Drug: Apixaban
  Arms: Diabetics (group 1); Nondiabetics (group 1)
Drug: Rivaroxaban
  Arms: Diabetics (group 1); Nondiabetics (group 1)
Drug: Edoxaban
  Arms: Diabetics (group 1); Nondiabetics (group 1)
Drug: Warfarin
  Arms: Diabetics (group 2); Nondiabetics (group 2)
Drug: Acenocumarole
  Arms: Diabetics (group 2); Nondiabetics (group 2)

SUMMARY:
Diabetic and nondiabetic patients will be evaluated if they had a first diagnosis of non-valvular atrial fibrillation and in therapy with non-vitamin K oral anticoagulants and with vitamin K oral anticoagulants.

DETAILED DESCRIPTION:
Parameters evaluated:

* anthropometric indices
* glycated haemoglobin, basal and postprandial glycemia
* lipid profile
* small and dense LDL; oxidized LDL
* I troponin
* red and white cells count; platelets count
* creatinin, transaminases, iron
* fibrinogen, D-dimer, anti-thrombin III
* Hs-CRP, metalloproteinases 2 and 9
* incidence of bleeding

ELIGIBILITY:
Inclusion Criteria:

* non-valvular atrial fibrillation
* nondiabetic patients
* type 1 and 2 diabetic patients

Exclusion Criteria:

* patients with cancer
* patients with chronic inflammation diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-09; Primary Completion 2019-04 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Efficacy on coagulation parameters | 12 months
  Red cells count
Efficacy on coagulation parameters | 12 months
  Platelets count
Efficacy on coagulation parameters | 12 months
  fibrinogen
Efficacy on coagulation parameters | 12 months
  D-dimer, anti-thrombin III

SECONDARY OUTCOMES:
Bleeding risk | 12 months
  HAS-BLED score
Inflammation parameters | 12 months
  Hs-CRP
Inflammation parameters | 12 months
  White cells count
Endothelial damage | 12 months
  Metalloproteinases 2 and 9
Oxidative status | 12 months
  Small and dense LDL; oxidized LDL
Heart damage | 12 months
  I troponin
Safety and tolerability parameters | 12 months
  Serum creatinin
Safety and tolerability parameters | 12 months
  Serum transaminases
Safety and tolerability parameters | 12 months
  Plasma iron

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Derosa, MD, PhD, FESC, Principal Investigator — University of Pavia and IRCCS Policlinico San Matteo
Locations (1):
- IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Derosa G, Rizzo M, Brunetti ND, Raddino R, Gavazzoni M, Pasini G, Gaudio G, Maggi A, D'Angelo A, De Gennaro L, Maffioli P. ORal anticoaGulants in diAbetic and Nondiabetic patients with nOn-valvular atrial fibrillatioN (ORGANON). J Diabetes Complications. 2023 Aug;37(8):108512. doi: 10.1016/j.jdiacomp.2023.108512. Epub 2023 May 20. PMID 37390799